CLINICAL TRIAL: NCT02440204
Title: Optimal Sevoflurane Concentration for Intubation Without Using Muscle Relaxants in Combination of Different Clinical Bolus Doses of Remifentanil
Brief Title: Optimal Sevoflurane Concentration for Intubation in Combination of Clincal Remifentanil Doses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Severance Hospital (Other)
Collaborators: Armed Forces Capital Hospital, Republic of Korea (Other Government)
Responsible Party: Principal Investigator, Dr. Koh, Jae Chul, MD, Fellow, Department of anesthesiology and pain medicine, Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AFMC-15036
Record Dates: First submitted 2015-05-05; First posted 2015-05-12 (Estimated); Results first posted 2019-01-17 (Actual); Last update posted 2019-01-17 (Actual); Status verified 2018-07

CONDITIONS: Postoperative Pain
Keywords: sevoflurane; remifentanil; intubation without using muscle relaxants
MeSH Terms: conditions — Pain, Postoperative | interventions — Intubation; Remifentanil; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Remifentanil 1.0 mcg/kg (Active Comparator): After setting the end-tidal sevoflurane concentration in a predetermined concentration, remifentanil will be injected according to their group and intubation will be performed 90 seconds after.
  Interventions: Procedure: Intubation; Drug: Remifentanil; Drug: Sevoflurane
- Remifentanil 1.5 mcg/kg (Active Comparator): After setting the end-tidal sevoflurane concentration in a predetermined concentration, remifentanil will be injected according to their group and intubation will be performed 90 seconds after.
  Interventions: Procedure: Intubation; Drug: Remifentanil; Drug: Sevoflurane
- Remifentanil 2.0 mcg/kg (Active Comparator): After setting the end-tidal sevoflurane concentration in a predetermined concentration, remifentanil will be injected according to their group and intubation will be performed 90 seconds after.
  Interventions: Procedure: Intubation; Drug: Remifentanil; Drug: Sevoflurane

INTERVENTIONS:
Procedure: Intubation — After setting the end-tidal sevoflurane concentration in a predetermined concentration, remifentanil will be injected according to their group and intubation will be performed 90 seconds after.
Drug: Remifentanil — After setting the end-tidal sevoflurane concentration in a predetermined concentration, remifentanil will be administered according to their group in 1 minute to prevent remifentanil induced rigidity or complications.
  Other Names: Ultiva
Drug: Sevoflurane — The end-tidal sevoflurane concentration will be set as predetermined, which starts from 2.5 vol% and adjusted by the up-and-down study model which have been described by Dixon JW et al.
  Other Names: Sevoran

SUMMARY:
Intubation is a procedure that requires well relaxed muscles while general anesthesia is performed. In order to get adequate muscle relaxation, remifentanil, sevoflurane or both agents in combination have been reported as they can provide adequate conditions for laryngoscopy and tracheal intubation without using muscle relaxants.

However, there were no previous studies to find the effective dose of sevoflurane in combination with different bolus doses of remifentanil to obtain adequate endotracheal intubation conditions without using muscle relaxants. The aim of this study is to investigate the change in the minimum sevoflurane alveolar concentration which produces an adequate endotracheal intubation condition when sevoflurane is combined with different bolus doses of remifentanil used in clinical practice.

DETAILED DESCRIPTION:
After Institutional Review Board approval and written informed consent, patients aged 18~30 years with American Society of Anesthesiologists physical status I or II who are scheduled to undergo elective otolaryngological surgery are enrolled in the study. Exclusion criterias are a history of reactive airway disease, smoking, a predictive signs of difficult intubation, and a body mass index ≥ 30 kg•m-2 or ≤ 15 kg•m-2. The patients will be assigned in 3 groups (group 1.0, 1.5, and 2.0) according to a computer-generated randomization table, to receive remifentanil bolus dose 1.0, 1.5 or 2.0 µg•kg-1, respectively.

Two anesthesiologists will participate in induction procedure in this study. One who is not blinded on patient's group or target sevoflurane concentration recorded the data, will adjust the dose of the sevoflurane and remifentanil and the other who is blinded will perform the mask ventilation and endotracheal intubation. Patients will be premedicated with glycopyrrolate 0.2 mg intravenously. An 18-gauge intravenous catheter will be established and 0.9% normal saline will be infused. In the operating room, all patients will be monitored with electrocardiogram, pulse oximetry, non-invasive blood pressure measurement, and measurement of both inspired and end-tidal concentration of oxygen, carbon dioxide and sevoflurane. After preoxygenation for 3 min, anesthesia is induced using a face mask with a semi-closed anesthetic circuit (Primus®, Dräger) prefilled with 8% sevoflurane for 10 min. The fresh gas flow will be set at 6 l•min-1. At first, patients will be left to breath spontaneously. However, when the tidal volume is too small to provide adequate end-tidal sampling for expiratory gas concentration measurement or end-tidal carbon dioxide level is above 40 mmHg, ventilation will be assisted. If the patient's spontaneous ventilation is disappeared, mechanical ventilation will be started with a tidal volume of 10 ml•kg-1, and respiratory rate will be adjusted to maintain end tidal carbon dioxide level between 35 mmHg and 40 mmHg. When the patient lost consciousness and the end-tidal sevoflurane level is higher than the preselected target concentration, the inspired concentration will be set 0 until the end-tidal concentration changed similar to the preselected target end-tidal sevoflurane concentration. Then the inspired concentration will be adjusted in a range of 1.0 to 1.4 times of the preselected sevoflurane level to find a concentration that can maintain preselected target end-tidal sevoflurane concentration steady for at least 3 min. The steady state end-tidal sevoflurane concentration will be maintained for 1 min. Even if the steady state concentration is found in less than 3 min, the remaining time will be added to this 1 min of steady state maintenance. After confirmation of the steady state, bolus dose of remifentanil will be administerd via intravenous line over 60 seconds to prevent chest wall rigidity according to the preselected group. 90 seconds after the end of remifentanil bolus administration, endotracheal intubation will be performed using a 7.5 mm (internal diameter) reinforced endotracheal tube. If the intubation condition is not good enough to perform an successful intubation, anesthesia will be deepened by increasing inspired sevoflurane concentration, and rocuronium 0.3 mg•kg-1 will be used to facilitate intubation.

The concentration of sevoflurane used for each patient will be determined by the response of the previously tested patient using the modified Dixon's up-and-down method[8]. The first patient will be tested at end-tidal sevoflurane concentration of 2.5%, which has been determined as a concentration for acceptable intubating condition in a previous study. According to a scoring system described by Helbo-Hansen S. et al., intubation condition will be scored. Successful intubation is defined as intubation under acceptable intubating condition by this scoring system. If intubation fails, the target concentration of sevoflurane will be increased by 0.5%. If intubation is successful, it will be decreased by 0.5%.

Statistical analyses will be performed using the statistical package SPSS 20.0 for windows (SPSS Inc., Chicago, IL). The sample size was determined to achieve seven response crossovers in each group to provide adequate minimum alveolar sevoflurane concentration defined as an average of response crossover midpoints. A response crossover is defined as an independent pair failure to success of intubation. To calculate the regression models allowing the prediction of the effective concentration of sevoflurane for successful intubation in 50%(ED50) and 95%(ED95) of the patients, a logistic regression analysis will be performed in each group. A repeated measures of ANOVA will be performed to compare hemodynamic data changes in each group. A p-value less than 0.05 is considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status I or II who were scheduled to undergo elective otolaryngological surgery

Exclusion Criteria:

* history of reactive airway disease
* smoking hx.
* a predictive signs of difficult intubation
* body mass index ≥ 30 kg•m-2 or ≤ 15 kg•m-2

Ages: 19 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2015-05; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eui-Kyoung Goo, MD, Study Director — Armed forces capital hospital
Locations (1):
- Armed Forces Capital Hospital, Republic of Korea, Seongnam-si, Kyung-ki Do, South Korea

REFERENCES:
- [Background] Cros AM, Lopez C, Kandel T, Sztark F. Determination of sevoflurane alveolar concentration for tracheal intubation with remifentanil, and no muscle relaxant. Anaesthesia. 2000 Oct;55(10):965-9. doi: 10.1046/j.1365-2044.2000.01538.x. PMID 11012491
- [Background] Min SK, Kwak YL, Park SY, Kim JS, Kim JY. The optimal dose of remifentanil for intubation during sevoflurane induction without neuromuscular blockade in children. Anaesthesia. 2007 May;62(5):446-50. doi: 10.1111/j.1365-2044.2007.05037.x. PMID 17448054
- [Result] Dixon WJ. Staircase bioassay: the up-and-down method. Neurosci Biobehav Rev. 1991 Spring;15(1):47-50. doi: 10.1016/s0149-7634(05)80090-9. PMID 2052197

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Remifentanil 1.0 mcg/kg | Remifentanil 1.5 mcg/kg | Remifentanil 2.0 mcg/kg
Started | 22 | 24 | 22
Completed | 22 | 24 | 22
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Remifentanil 1.0 mcg/kg | Remifentanil 1.5 mcg/kg | Remifentanil 2.0 mcg/kg | Total
Number analyzed (Participants) | 22 | 24 | 22 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 22 | 24 | 22 | 68
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.3 (1.7) | 21.3 (1.6) | 21.5 (2.2) | 21.3 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 22 | 24 | 22 | 68
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  South Korea | 22 | 24 | 22 | 68

OUTCOME MEASURES:

1. Primary Outcome: EC50 for Successful Intubation in Each Groups
Description: Sevoflurane concentration used to perform intubation (For ED50 finding)
Time Frame: During the induction of anesthesia
Measure: Mean (95% Confidence Interval); unit: vol%
Arm/Group | Remifentanil 1.0 mcg/kg | Remifentanil 1.5 mcg/kg | Remifentanil 2.0 mcg/kg
Number analyzed (Participants) | 22 | 24 | 22
vol% | 3.00 [2.36 to 3.18] | 2.00 [1.38 to 2.54] | 1.29 [1.14 to 1.50]

2. Secondary Outcome: EC95 for Successful Intubation
Description: Sevoflurane concentration used to perform intubation (For ED95 finding)
Time Frame: During the induction of anesthesia
Measure: Mean (95% Confidence Interval); unit: vol%
Arm/Group | Remifentanil 1.0 mcg/kg | Remifentanil 1.5 mcg/kg | Remifentanil 2.0 mcg/kg
Number analyzed (Participants) | 22 | 24 | 22
vol% | 3.45 [3.00 to 3.47] | 2.91 [2.35 to 2.95] | 1.89 [1.47 to 1.95]

ADVERSE EVENTS:
Arm/Group | Remifentanil 1.0 mcg/kg | Remifentanil 1.5 mcg/kg | Remifentanil 2.0 mcg/kg
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/24 | 0/22
Other Adverse Events (participants affected / at risk) | 1/22 | 2/24 | 6/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Remifentanil 1.0 mcg/kg (N=22) | Remifentanil 1.5 mcg/kg (N=24) | Remifentanil 2.0 mcg/kg (N=22)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 3 (3)
Closed vocal cords (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes